CLINICAL TRIAL: NCT03677843
Title: Multidimensional Approach in Patients With Severe Cerebral Palsy, Prospective Cohort(MAPCP Cohort)-Offline
Status: Recruiting | Type: Observational
Sponsor: Ju Seok Ryu (Other)
Responsible Party: Sponsor-Investigator, Ju Seok Ryu, Associate Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: B-1808/484-302
Record Dates: First submitted 2018-09-10; First posted 2018-09-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy, Spastic
Keywords: hip dislocation; GMFCS level 3,4,5; scoliosis
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cerebral palsy: They are included in GMFCS level 3, 4, 5. and they have diplegia or quadriplegia

SUMMARY:
In children with cerebral palsy, secondary problems lead to hip dislocation and scoliosis. But There is no definite evidence for the dislocation of hip and scoliosis. The investigators want to verify evidence of scoliosis and dislocation of hip.

DETAILED DESCRIPTION:
Observation cohort study. The investigators will measure for finding evidence by checking the x-ray photograph, hip adductor muscles pressure test and electromyography(EMG test) test of hip adductor and spine muscles

ELIGIBILITY:
Inclusion Criteria:

* Severe cerebral palsy patients(GMFCS level 3,4,5)
* 2 to 10 years old

Exclusion Criteria:

* Those who disagree with the study.
* other than cerebral palsy.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Serious cerebral palsy children(GMFCS 3,4,5) have secondary problems such as hip dislocation and scoliosis. and There are many preliminary reports that hip dislocation occurs from 2 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
hip adductor and spin muscles electromyography(EMG) test | once at study, when patient enrolled
  Use EMG to check the activity of the hip adductor and spine muscles of participants.
  This figures will give investigators a look at the association with a hip dislocation.

SECONDARY OUTCOMES:
Whole spine AP and total Hip AP X-ray photograph | once at study, when patient enrolled and after once every six months for three years
  Whole spine and total Hip joint are checked with X-ray photograph. and investigators will check the progress of hip dislocation and spinal scoliosis.
hip adductor muscles pressure meter test | once at study, when patient enrolled
  Pressures of hip adductors muscles are measured from pressure meter. and This figures will give investigators a look at the association with a hip dislocation.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided